CLINICAL TRIAL: NCT01091272
Title: A Phase 1, First-Into-Human, Escalating Dose Trial To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-04995274 After Administration Of Single Oral Doses To Healthy Adult Subjects
Brief Title: A Study To Evaluate The Safety, Tolerability And Plasma Drug Levels Following A Single Dose Of PF-04995274 In Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B1661001
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: healthy volunteer; safety; pharmacokinetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Single dose 3 period interleaved cross-over with placebo substitution
  Interventions: Drug: PF-04995274
- Cohort 2 (Experimental): Single dose 4 period interleaved cross-over, placebo substitution, with food effect
  Interventions: Drug: PF-04995274
- Cohort 3 (Experimental): Single dose 4 period cross-over, placebo insertion, with food effect
  Interventions: Drug: PF-04995274
- Optional Cohort 4 (Experimental): Single dose 3 period cross-over with placebo substitution
  Interventions: Drug: PF-04995274

INTERVENTIONS:
Drug: PF-04995274 — Planned single PO 0.15mg, 1.5mg, 15mg doses of PF-04995274 interleaved with cohort 2 such that doses escalate from 0.15 mg to 50 mg.
  Arms: Cohort 1
Drug: PF-04995274 — Planned single PO 0.5mg, 5mg, 50mg doses of PF-04995274, interleaved with cohort 2 such that doses escalate from 0.15 mg to 50 mg interleaved with cohort 2 such that doses escalate from 0.15 mg to 50 mg.
  Arms: Cohort 2
Drug: PF-04995274 — Planned single PO 120mg and 210mg doses of PF-04995274
  Arms: Cohort 3
Drug: PF-04995274 — single PO dose of PF-04995274; dosage to be determined by safety and pharmacokinetic data
  Arms: Optional Cohort 4

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of PF-04995274 after administration of a single dose to healthy volunteers, and to evaluate the plasma drug concentrations after single dose in healthy volunteers.

DETAILED DESCRIPTION:
The purpose is to evaluate the safety and pharmacokinetics of a single dose of PF-04995274 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* For all cohorts, healthy male and/or female subjects of nonchildbearing potential between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12 lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Pregnant or nursing women; women of childbearing potential. Female subjects must be of non childbearing potential defined by a history of surgical sterilization (eg, hysterectomy or bilateral oophorectomy) or post menopausal status (complete absence of menses for at least two consecutive years) and elevated FSH concentration in women between 45 and 55.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety Endpoints (AE's, Vital signs (supine & standing BP, PR), Triplicate ECG, 8 hours of cardiac telemetry postdose, Clinical safety laboratory endpoints, Digit Symbol Substitution Test (DSST), Drug Effect Questionnaire (DEQ), Clinical | up to 21 days post dose
examinations) | up to 21 days post dose
Cmax, Tmax, AUClast, AUCinf, and t1/2 of PF 04995274, as the data permit. | up to 7 days post dose
Cmax, Tmax, AUClast, AUCinf, and t1/2 of PF 05082547, as the data permit. | up to 7 days post dosing

SECONDARY OUTCOMES:
Plasma aldosterone concentrations | through 1 day post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1661001&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%20And%20Plasma%20Drug%20Levels%20Following%20A%20Single%20Dose%20Of%20PF-04995274%20In%20Healthy%20Adult%20Voluntee